CLINICAL TRIAL: NCT01516112
Title: Meir Medical Center Home Monitoring Clinic Registry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Hospital, Kfar Saba, Israel (Other)
Responsible Party: Principal Investigator, chetboun israel, Dr. Israel Chetboun, Meir Hospital, Kfar Saba, Israel
Other Study IDs: HMR-1.0-MEIR
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2011-07

CONDITIONS: Patients Implanted With an ICD or CRTD.
Keywords: ICD, home monitoring, cardiomessenger, implant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the registry is to assess workload of a Home Monitoring based follow up for Biotronik ICD and CRTD patients.

ELIGIBILITY:
Inclusion Criteria:

* Approved indication for ICD or CRTD
* Implanted with or replaced with a Biotronik Lumax device
* Patient willing and able to sign consent form
* Willing and able to attend clinic visits and follow up schedule
* Transmission of more than 80% at 3-month follow up
* Patient older than 18 years

Exclusion Criteria:

* no indication for ICD or CRTD implant
* Life expectancy shorter than 12 months
* Pregnancy
* Participation in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with an ICD or CRTD.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-02

CONTACTS AND LOCATIONS:
Locations (1):
- Meir MC, Kfar Saba, Israel